CLINICAL TRIAL: NCT00239785
Title: A One-year, Multicenter, Partially Blinded, Double-dummy, Randomized Study to Evaluate the Efficacy and Safety of FTY720 Combined With Reduced-dose or Full-dose Cyclosporine, USP [Modified] (Novartis Brand) and Corticosteroids Versus Mycophenolate Mofetil Combined With Full-dose Cyclosporine, USP [Modified] (Novartis Brand) and Corticosteroids, in de Novo Adult Renal Transplant Recipients
Brief Title: Efficacy and Safety of FTY720 in de Novo Adult Renal Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFTY720A0124
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Renal Transplantation
Keywords: Transplantation, kidney, and organ transplant.
MeSH Terms: interventions — Fingolimod Hydrochloride

INTERVENTIONS:
Drug: FTY720

SUMMARY:
This study will evaluate the safety and efficacy of FTY720 combined with cyclosporine and corticosteroids in patients receiving a kidney organ transplant

ELIGIBILITY:
Inclusion Criteria

* Male and female patients of any race between 18 to 65 years old (inclusive)
* Patients scheduled to undergo a primary cadaveric or primary non-HLA identical living donor kidney transplantation
* Patients who gave written informed consent to participate in the study Exclusion Criteria
* Recipients of multi-organ transplantation or foreseen to receive a non-renal allograft during the study period
* Graft cold ischemia time greater than 40 hours.
* Patients with pulse rate < 50 beats per minute (bpm) at screening Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 684
Dates: Start 2003-04; Primary Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
IA, IB, IIA, IIB, III, or humoral rejection diagnosed by biopsy according to Banff 97 criteria within 12 months post transplant
Permanent resumption of dialysis within 12 months post transplant
Surgical removal of graft within 12 months post transplant
Death within 12 months post transplant
Withdrawal of consent, death, or lost to follow up within 12 months post transplant

SECONDARY OUTCOMES:
FEV1 , FVC, FEV1/FVC, DLCO and FEF 25%-75% at day 28, months 6 and 12
Serum creatinine
Cystatin C at months 3, 6, and 12
Proteinuria at day 28, months 6 and 12
Absolute lymphocyte count at screening, baseline, day 1, 7, 14, and 28, months 2, 3, 6, 9, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis